CLINICAL TRIAL: NCT03027739
Title: CART-19 Cells For Patients With Minimal Residual Disease (MRD) Positive CD19+ Acute Lymphoblastic Leukemia
Brief Title: CART-19 Cells For MRD Positive CD19+ ALL
Acronym: CCFMPCA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Jianda Hu, Director of the department of Hematology, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-19-02
Record Dates: First submitted 2017-01-17; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — CTL019 chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): CART-19 cells treated
  Interventions: Biological: CART-19

INTERVENTIONS:
Biological: CART-19 — CART-19 cells treated

SUMMARY:
CART-19 cells has emerged as a powerful targeted immunotherapy, showing striking responses in highly refractory CD19+ acute lymphoblastic leukemia (ALL). This study aims to assess the safety and toxicity of CART-19 cells to patients who are refractory or at highest risk of relapse as defined by MRD+ status.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Aged between 1-60 years
* Patients with MRD positive CD19+ ALL
* Cardiac: Left ventricular ejection fraction ≥ 50%
* Adequate renal and hepatic function
* Performance status: Karnofsky ≥ 70%

Exclusion Criteria:

* Pregnant or lactating females.
* Any co-morbidity precluding the administration of CART-19 cells.

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Leukemia free survival | 1 year

SECONDARY OUTCOMES:
Adverse events that are related to treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jianda Hu, 86-13959169016, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No